CLINICAL TRIAL: NCT06104657
Title: Qualitative Techniques to Define Meaningful Within-Patient Change in Symptoms of Advanced Cancer Patients
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-012283; NCI-2023-00315 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-012283 (Other: Mayo Clinic in Rochester); FD 05938 (Other Grant/Funding Number: Food and Drug Administration)
Record Dates: First submitted 2023-10-20; First posted 2023-10-27 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational Patient Group: Patients take part in interview on study.
  Interventions: Other: Non-Interventional Study
- Observational Patient Advocate Group: Patient advocate participants take part in an interview on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study examines qualitative techniques in defining meaningful within patients changes in symptoms in patients with cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). This study may help researcher better understand how to interpret reports from patients about their cancer symptoms and treatment side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop method to establish meaningful change in patient-reported outcomes (PROs).

II. To provide responder definitions in 2 ways:

IIa: Detectable change: within patient score change patients perceive but does not exceed a subjective threshold for a modification to patient care (for worsening) or conclusion of achieving therapeutic benefit (for improvement); IIb. Meaningful change: within patient score change that patients perceive and that does require modification in management (for worsening) or supports conclusion of therapeutic benefit (improvement).

OUTLINE: This is an observational study. Participants are assigned to 1 of 2 groups.

PATIENTS: Patients take part in an interview on study.

PATIENT ADVOCATES: Patient advocate participants take part in an interview on study.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS

  * Patients with a diagnosis of cancer including solid tumor and hematologic malignancy at Mayo Clinic, Rochester
  * To ensure sampling patients likely to have experienced declines in fatigue, all patients will have had at least two in-person encounters for radiation or chemotherapy treatment within the 3 months prior to recruitment. The sampling methodology developed for the Consumer Assessment of Healthcare Providers and Systems (CAHPS) Cancer Care survey will be modified and used to identify eligible patients from Mayo Clinic's electronic health record
  * As interviews will be conducted either in person or by video conference (Zoom, Teams, or similar), access to internet is required for those unable or unwilling to travel to the clinic for an in-person interview
  * Answered "Yes" to screening question: "In the past 3 months, have you experienced changes in your level of fatigue?" Yes/No
* PATIENT ADVOCATES:

  * Patient advocates recommended by the FDA to provide their input to help us in reaching a consensus in the way we define meaningful change (both improvement and decline) that came from patients in the first arm

Exclusion Criteria:

* PATIENTS

  * Unwilling to be audio recorded during the interviews
  * Answered "No" for the screening question

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumor and hematologic malignancy at Mayo Clinic, as well as patient advocates
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Meaningful change in patient reported outcomes (PROs) | Baseline
  Change in PROs will be assessed using the critical incident technique (CIT) during semi-structured interviews as a means of educating, training, and evaluating patients on the concept of meaningful change. Interviews will be summarized to record how patients explain the concept of meaningful improvement and declines in their own words.
Change in Patient Reported Outcome - Common Terminology Criteria for Adverse Events (PRO-CTCAE) scores | Baseline
  PRO-CTCAE is a patient-reported outcome (PRO) measurement system developed to evaluate symptomatic toxicity in patients on cancer clinical trials. It was designed to be used as a companion to the Common Terminology Criteria for Adverse Events (CTCAE). Scores will be evaluated for worsening from good days (baseline) and improvement from bad days (baseline).
Change in Functional Assessment of Cancer Therapy - General (FACT-G) scores | Baseline
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire that measures four domains of Health-Related Quality of Life (HRQOL) in cancer patients: physical, social, emotional, and functional well-being. Questions are answered with a 0-4 scale where 0=Not at all and 4=Very much. Scores will be evaluated for worsening from good days (baseline) and improvement from bad days (baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Minji K. Lee, Ph.D., M.S., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials